CLINICAL TRIAL: NCT04511767
Title: Reliability and Validity of Child-Caregiver Interaction Observation Scale (CCIOS) for Diagnosis of Autism Spectrum Disorder
Brief Title: Reliability and Validity of CCISO for Diagnosis of Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CCIOS2020
Record Dates: First submitted 2020-08-02; First posted 2020-08-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-11

CONDITIONS: Autism Spectrum Disorder; Global Developmental Delay; Language Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities; Language Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ASD group: the autism spectrum disorder group
  Interventions: Other: Do not take any interventions
- GDD group: the global developmental disorder group
  Interventions: Other: Do not take any interventions
- LD group: the language disorder group
  Interventions: Other: Do not take any interventions

INTERVENTIONS:
Other: Do not take any interventions — Do not take any interventions

SUMMARY:
The investigators designed the Child-Caregiver Interaction Observation Scale（CCIOS）to assess social communication behaviors, stereotyped behaviors for children with autism spectrum disorder(ASD) via a 20-min video of interactions between a caregiver and a child. The original CCIOS coding scheme consists 23 items. The score range for each item is 0-4, with higher scores being indicative of more atypical behavior. The aim of the study is to determine items for inclusion in the final CCIOS coding scheme through exploration of item correlations, establish the cutoff score of CCIOS for ASD and evaluate the reliability and validity of CCIOS. The reliability evaluation include test-retest reliability and inter-rater reliability. DSM-5 criterion is used as the gold standard. Validity is assessed by determining the correlation and consistency between CCIOS and DSM-5 criterion.

DETAILED DESCRIPTION:
The investigators designed the Child-Caregiver Interaction Observation Scale（CCIOS）to assess social communication behaviors, stereotyped behaviors for children with autism spectrum disorder(ASD) via a 20-min video of interactions between a caregiver and a child. The original CCIOS coding scheme consists 23 items. The score range for each item is 0-4, with higher scores being indicative of more atypical behavior. The investigators conduct this study to determine items for inclusion in the final CCIOS coding scheme through exploration of item correlations, establish the cutoff score of CCIOS for ASD and evaluate the reliability and validity of CCIOS.

It is of importance to accurately distinguish children with ASD from those with Global Developmental Delay (GDD) and Language Disorder (LD) without ASD, sometimes, it's very difficult in children with mental ages below 2 years. This differentiation has strong implications for treatment recommendations and may also inform long-term prognosis. In this study, The investigators planned to recruit 60 children with ASD and 60 children with GDD/LD aged from 18 months to 48 months. The reliability evaluation include test-retest reliability and inter-rater reliability. DSM-5 criterion is used as the gold standard. Validity is assessed by determining the correlation and consistency between CCIOS and DSM-5 criterion.

ELIGIBILITY:
Inclusion Criteria:

* The ASD/GDD/LD diagnosis is made based on the criteria of ASD/GDD/LD in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) ;
* Age 18 months - 48 months;

Exclusion Criteria:

* Visual, audi-tory and physical disabilities

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ASD/GDD/LD children are from development behavior clinic
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
The scores of CCSIO for ASD/GDD/ID children | At enrollment
  CCIOS coding scheme is a 5-point rating scale (0 to 4), with higher scores being indicative of more atypical behavior. The total score can be got by adding up the score of each item.

SECONDARY OUTCOMES:
The scores of CCSIO for ASD/GDD/ID children (One quarter) | At 1 month after enrollment
  One quarter of subjects will be selected randomly at 1 month after entering the study and take the CCIOS measurement again. CCIOS coding scheme is a 5-point rating scale (0 to 4), with higher scores being indicative of more atypical behavior. The total score can be got by adding up the score of each item.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Xu, Doctor, Principal Investigator — Children's Hospital of Fudan University; Qiong Xu, Doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China